CLINICAL TRIAL: NCT07294443
Title: The Effect of Qigong Relaxation Exercise on Anxiety and Depression Levels in Individuals Diagnosed With Depression Hospitalized in a Psychiatric Clinic
Brief Title: Qigong Relaxation Exercise
Acronym: QRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Aydan Akkurt Yalçıntürk, Asst. Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 61351342
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Qigong; Anxiety; Depression; Psychiatric Disorders; Relaxation
MeSH Terms: conditions — Anxiety Disorders; Depression; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QRE (Experimental)
  Interventions: Other: Qigong relaxation exercises
- Control group (Active Comparator)
  Interventions: Other: Ongoing treatment

INTERVENTIONS:
Other: Qigong relaxation exercises — Qigong relaxation exercise is a type of exercise consisting of graceful body movements and relaxation, performed in harmony with breathing and meditation, aimed at relaxing the body and mind, reducing stress, diverting attention away from negative thoughts, accelerating blood flow, and improving emotions.
  Arms: QRE
Other: Ongoing treatment — The control group's ongoing treatment continued.
  Arms: Control group

SUMMARY:
Objective: This study was conducted to examine the effect of Qigong relaxation exercises applied in a psychiatric clinic on the anxiety and depression levels of patients diagnosed with depression.

Design: This study was designed as a single-blind, randomized controlled trial. Research Hypotheses H1: State anxiety levels are lower in patients who perform Qigong exercises than in those who do not.

H2: Depression levels are lower in patients who perform Qigong exercises than in those who do not.

The study population consisted of 140 individuals aged 18 years and older diagnosed with depression who were hospitalized at a private psychiatric hospital in Turkey between March 1 and September 1, 2025. In the sample selection, the STAI-I and Beck Depression Scale were administered to the patients by the researchers. Since differences in anxiety and depression levels would affect group homogeneity, patients who scored below 35 on the STAI-I (mild and moderate levels) and between 17 and 30 on the Beck Depression Scale constituted the study sample. The study sample consisted of 70 patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient is literate
* No communication barriers
* The patient is receiving inpatient treatment at a psychiatric clinic
* The patient has been diagnosed with depression
* The patient is over 18 years of age
* The patient is oriented to the service (at least 24 hours have passed since admission)
* The patient regularly participates in Qigong practice

Exclusion Criteria:

* The patient has communication difficulties
* The patient has acute psychotic symptoms
* The patient is receiving anxiolytic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Beck Depression Scale | 6 weeks
  Beck Depression Scale: The Beck Depression Scale was used to measure the level and severity of depressive symptoms. The Beck Depression Scale, which underwent a Turkish validity and reliability study by Hisli in 1988, is a depression rating scale consisting of 21 questions. Individuals mark the statement that best describes how they have felt over the past 15 days, and the total score is calculated by summing the points (0-3) obtained from each response. According to the corresponding score ranges, the scale is evaluated as follows: 1-10 is normal, 11-16 is moderate mood disorder, 17-20 is clinical depression, 21-30 is moderate depression, 31-40 is severe depression, and 41-63 is major depression.
State-Trait Anxiety Inventory | 6 weeks
  This scale was developed by Spielberger et al. (1983), and its validity and reliability in Turkish were established by Öner and Le Compte (1985). The scale consists of two parts: the State Anxiety Scale (STAI-I) and the Trait Anxiety Scale (STAI-II). STAI-I examines how an individual feels at a specific time and under specific conditions, while STAI-II determines how an individual feels independently of the situation and conditions they are in. STAI-I form, which consists of 20 statements, was used to measure state anxiety. Respondents rated their level of anxiety on a 4-point (1- 4) intensity scale from not at all tovery much so.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University, Istanbul, Üsküdar - Selimiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No